CLINICAL TRIAL: NCT03076580
Title: An Integrative-omics Study to Identify New Biomarkers of Cardiomyopathy Patients in China
Brief Title: An Integrative-"Omics" Study of Cardiomyopathy Patients for Diagnosis and Prognosis in China
Acronym: AOCC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Institute of Heart, Lung and Blood Vessel Diseases (Other)
Collaborators: Chinese Academy of Medical Sciences, Fuwai Hospital (Other); Beijing Anzhen Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: BeijingIHLBVD2016031
Record Dates: First submitted 2017-03-01; First posted 2017-03-10 (Actual); Last update posted 2018-04-19 (Actual); Status verified 2017-03

CONDITIONS: Dilated Cardiomyopathy; Hypertrophic Cardiomyopathy; Arrhythmogenic Right Ventricular Cardiomyopathy; Left Ventricular Non-compaction; Restrictive Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathy, Dilated; Cardiomyopathy, Hypertrophic; Arrhythmogenic Right Ventricular Dysplasia; Cardiomyopathy, Restrictive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — If a blood specimen is obtained, it will be separated and stored at -80 ℃ as plasma, viable cells, and extracted DNA. If a saliva specimen is obtained, it is stored for DNA. If a tissue specimen is obtained, it will be cut into small pieces and stored at liquid nitrogen.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- cardiomyopathy: Patients are diagnosed as cardiomyopathy by three cardiologists and recruited in Beijing Anzhen Hospital, recording the results of clinical lab and echocardiography.
- disease control: Patients have similar symptoms with cardiomyopathy patients, and are further excluded by three cardiologists and recruited in Beijing Anzhen Hospital, recording the results of clinical lab and echocardiography.
- healthy control: Healthy subjects are recruited in Beijing Anzhen Hospital, with negative results of echocardiography and clinical lab examination.

SUMMARY:
This is a multi-omics research of Chinese cardiomyopathies patients, aiming to determine genetic risk factor and serial biomarkers of cardiomyopathies in diagnosis and prognosis.

DETAILED DESCRIPTION:
Identification of novel biomarkers is needed to improve the diagnosis and prognosis of cardiomyopathy. Also,the marked variation of genes which is still unclear, may influence clinical outcomes is determined in part by genetic heterogeneity of the systemic response to pathological process.

Specific aim:

1. Proteomics, microRNA-seq and metabolomics will be to determine the correlation of echocardiographic parameters of systolic and diastolic functional entry with circulating molecules
2. Genomics will be to determine the association of clinical outcome

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who was diagnosed as cardiomyopathy by medical history, clinical symptoms, laboratory tests including ECG, echocardiography.
2. Subject understands study requirements aand agrees to sign an informed consent form prior to any study procedures.

Exclusion Criteria:

1. Endocrine disease known to cause heart muscle disease (including infants of diabetic mothers)
2. History of rheumatic fever
3. Toxic exposures known to cause heart muscle disease (anthracyclines, mediastinal radiation, iron overload or heavy metal exposure)
4. HIV infection or born to an HIV positive mother
5. Kawasaki disease
6. Immunologic disease
7. Uremia, active or chronic
8. Abnormal ventricular size or function that can be attributed to intense 9.physical training or chronic anemia

10.Chronic arrhythmia, unless there are studies documenting inclusion criteria prior to the onset of arrhythmia (except a patient with chronic arrhythmia, subsequently ablated, whose cardiomyopathy persists after two months is not to be excluded) 11.Malignancy 12.Pulmonary parenchymal or vascular disease (e.g., cystic fibrosis, cor pulmonale, or pulmonary hypertension) 13.Ischemic coronary vascular disease 14.Association with drugs (e.g., growth hormone, corticosteroids, cocaine) or other diseases known to cause hypertrophy

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: A diagnosis of cardiomyopaty is adjudicated by three cardiologists,according to current guidelines when there was clinical evidence of cardiomyopathy together with clinical symptoms of heart failure or echocardiography or imaging evidence.
  Patients have smiliar symptoms and are suspected as cardiomyopathy and further excluded by imaging examnation.
  age- and gender- mathced healthy controls are also recuitted in the hospital.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2015-07-01 (Actual); Primary Completion 2018-07-01 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
The primary objective of this study is to determine whether variation in genetic background or differentially expressed molecules influences clinical outcomes in cardiomyopathy. | Five year
  The primary objective of this study is to determine whether variation in genetic background or molecules influences clinical outcomes in cardiomyopathy. Differentially expressed molecules are reported in multi-omics.

SECONDARY OUTCOMES:
Age for each participant | These data is collected from the cases' medical record in an average of 1 month after the sample recruiting
gender for each participant | These data is collected from the cases' medical record in an average of 1 month after the sample recruiting
Height for each participant | These data is collected from the cases' medical record in an average of 1 month after the sample recruiting
Weight for each participant | These data is collected from the cases' medical record in an average of 1 month after the sample recruiting
Past medical history for each participant including disease history, surgical history, and family | These data is collected from the cases' medical record in an average of 1 month after the sample recruiting
Life style for each participant including smoking history and drinking, specify how many years | These data is collected from the cases' medical record in an average of 1 month after the sample recruiting
blood lipids(LDL,HDL,VLDL) | These data is collected from the cases' medical record in an average of 1 month after the sample recruiting
creatine | These data is collected from the cases' medical record in an average of 1 month after the sample recruiting
urea | These data is collected from the cases' medical record in an average of 1 month after the sample recruiting
blood glucose | These data is collected from the cases' medical record in an average of 1 month after the sample recruiting
D-dimer | These data is collected from the cases' medical record in an average of 1 month after the sample recruiting
hsCRP | These data is collected from the cases' medical record in an average of 1 month after the sample recruiting
All-cause death | One year/Three year/Five year
  The data is collected during follow-up visit at 1/3/5 years after discharge
Re-hospitalization | One year/Three year/Five year
  Patients are hospitalized due to heart failure with decreasing left ventricular ejection fraction or worsen symptoms. The data is collected during follow-up visit at 1/3/5 years after discharge
Heart transplantation | One year/Three year/Five year
  Patients are underwent heart transplantation due to "pump failure of heart".The data is collected during follow-up visit at 1/3 years after discharge
Malignant arrythmia | One year/Three year/Five year
  Ventricular flutter and fibrillation, atrioventricular block,atrial fibrillation or other cardiac arrhythmia leads to syncope or should be Implantable Cardioverter-Defibrillator (ICD) implantation.
Worsening heart failure | One year/Three year/Five year
  Worsen heart failure is defined as decreased ejection fraction(left ventricular ejection fraction decreased over 10%), left ventricular ejection fraction <45% and enlarged heart size measured by echocardiography and changing level of New York Heart Association (NYHA) Functional Classification.And patients who undergo left ventricular assist device (LVAD) will also be included.The data is collected during follow-up visit at 3/6/9/12/36/60 months after enrollment.
RNA/micro RNA/long-noncoding RNA-sequencing data | The data is collected from lab in an average of 6 month after the sample recruiting
Proteomics on Liquid Chromatograph Mass Spectrometer/Mass Spectrometer of plasma sample | The data is collected from lab in an average of 6 month after the sample recruiting
Exon sequencing data | The data is collected from lab in an average of 6 month after the sample recruiting
Result of echocardiography-Ejection Fraction | Three year
  The whole results of echocardiography report will be recorded. The indicate can reflect cardiac contraction function and be used for discriminating heart failure or non-heart failure as a main factor.
Result of echocardiography-Left Ventricular End Diastolic Diameter | Three year
  The whole results of echocardiography report will be recorded. The indicate can reflect the size of heart and be used for determination of heart enlargement.
Result of echocardiography-E/A Ratio | Three year
  The whole results of echocardiography report will be recorded. The indicate can reflect diastolic function.

CONTACTS AND LOCATIONS:
Overall Officials: Jie Du, PhD, Study Chair — Beijing Anzhen Hospital Affiliated to Capital Medical University
Locations (2):
- China (2):
  - Beijing Institute of heart, lung and blood vessel diseases, Beijing, Beijing Municipality
  - Shijie You, Beijing

IPD SHARING:
Plan to Share IPD: Undecided